CLINICAL TRIAL: NCT04678427
Title: TEAM Me (Totally Excited About Moving, Mobility, and Exercise) Clinical Research Protocol
Brief Title: Exercise Program (TEAM Me) for the Improvement of Movement and Mobility in Pediatric and Adolescent and Young Adult Patients With Cancer Undergoing a Blood Stem Cell Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0044; NCI-2020-11750 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0044 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (TEAM Me) (Experimental): Patients complete a 6-minute walk test and a timed get up and go test on the day of hospital admission, on days 0 (day of stem cell transplant) and 21, the day of discharge, and day 100. Patients also complete surveys over 10 minutes about quality of life and fatigue levels on the day of hospital admission, on days 0 (day of stem cell transplant) and 21, the day of discharge, and day 100. Patients who are able and allowed to, may also walk and participate in other intense physical activities to earn stickers. Patients who are unable to walk have tailored goals created by a physical/occupational therapist to earn stickers and participate in physical activity as prescribed by their therapist.
  Interventions: Other: 6 Minute Walk Functional Test; Behavioral: Behavioral Intervention; Other: Survey Administration; Behavioral: Timed Get Up and Go Test

INTERVENTIONS:
Other: 6 Minute Walk Functional Test — Complete 6-minute walk test
  Other Names: 6MWT; SIX MINUTE WALK; SIXMW1
Behavioral: Behavioral Intervention — Participate in walking and other activities
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Survey Administration — Complete survey
Behavioral: Timed Get Up and Go Test — Complete timed get up and go test

SUMMARY:
This clinical trial studies how well an exercise program (Totally Excited About Moving, Mobility, and Exercise [TEAM Me]) affects the exercise and dietary habits of pediatric and adolescents and young adults with cancer undergoing a blood stem cell transplant. TEAM Me is an exercise program that reinforces behavior, such as walking and other activities, using "tokens" (i.e. stickers) that can be redeemed for rewards. Participating in the exercise program may result in increased physical fitness, physical activity level, quality of life, and function in pediatric and adolescents and young adult patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility and tolerability of this exercise program using a token economy system in hospitalized pediatric and adolescent and young adult (AYA) undergoing hematopoietic stem cell transplant (HSCT).

SECONDARY OBJECTIVES:

I. To evaluate the impact of an exercise program using a token economy system in hospitalized pediatric and adolescent and young adult (AYA) cancer patients going through HSCT on measures of physical fitness.

II. To evaluate the impact of an exercise program using a token economy system in hospitalized pediatric and adolescent and young adult (AYA) cancer patients going through HSCT on physical activity.

III. To evaluate the impact of an exercise program using a token economy system in hospitalized pediatric and adolescent and young adult (AYA) cancer patients on quality of life, fatigue, sleep and function.

OUTLINE:

Patients complete a 6-minute walk test and a timed get up and go test on the day of hospital admission, on days 0 (day of stem cell transplant) and 21, the day of discharge, and day 100. Patients also complete surveys over 10 minutes about quality of life and fatigue levels on the day of hospital admission, on days 0 (day of stem cell transplant) and 21, the day of discharge, and day 100. Patients who are able and allowed to, may also walk and participate in other intense physical activities to earn stickers. Patients who are unable to walk have tailored goals created by a physical/occupational therapist to earn stickers and participate in physical activity as prescribed by their therapist.

ELIGIBILITY:
Inclusion Criteria:

* Be admitted to an inpatient pediatric ward for the purpose of HSCT for the treatment of malignancy
* Be greater than or equal to 6 years of age and less than 30 years of age
* Participants or guardians are willing and able to give written informed consent either prior to admission or within 48 hours following admission and to comply with all of the study activities and procedures
* Participants or guardians are willing and able to give written informed consent for protocol PA18-0130 (Pediatric Energy balance data repository protocol), companion protocol for the Fitbit application/assessment

Exclusion Criteria:

* Patients whose clinical status precludes them from participating in any physical activity including but not limited to: declining respiratory status, hypoxia requiring high flow nasal cannula (Vapotherm), hypotension, and active bleeding.
* At MD Anderson HSCT patients admitted to adult units for their transplant will not be eligible as TEAM Me is an established program on the G9 Pediatrics Unit only

Ages: 6 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who enroll and complete the serial measures | Up to 21 days post-hematopoietic stem cell transplant (HSCT)
  Will consider the program feasible if 75% of patients approached about the study will agree to enroll and 80% of the enrolled subjects will participate in physical activity and complete the serial measures for 70% of their inpatient days until day +21. Will report the percentage with 95% confidence interval of approached patients that agree to participate at the end of the study. Each patient's percentage of days that he/she complete the serial measures until day +21 will be calculated and percentage of all patients that finish 70% of the 21 day serial measures will be estimated with 95% confidence interval.
Incidence of adverse events. | Up to 100 days post-HSCT
  The program will be considered tolerable if > 90% of the participants do not have any Common Terminology Criteria for Adverse Events defined adverse events that are greater than grade 2. Serious adverse event will be defined using Common Terminology Criteria for Adverse Events version 5.0 or higher.

SECONDARY OUTCOMES:
Change in 6-minute walking test (6MWT) | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in gross grip hand strength | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in timed up and go test | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in Borg Rating of Perceived Exertion | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in 30 second sit-to-stand test | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in Fitbit mileage and intensity via heart rate | Baseline up to 100 days post-HSCT
  Will be recorded thru their co-enrollment on MD Anderson Cancer Center protocol PA18-0130. Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in PedsQL Stem Cell Transplant Model | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.
Change in Wee Functional Independence Measure (FIM)/FIM | Baseline up to 100 days post-HSCT
  Will be estimated from descriptive statistics: mean, standard deviation, median and range for each group and be compared using Wilcoxon rank sum test when appropriate. Baseline will be defined as the initial measures conducted at time of admission. Wilcoxon signed rank test may also be applied to test any change that is significantly different from 0. Repeated measure analysis may be applied to evaluate the changes of this measure over time, correlation between this scale and the 6MWT, adjusting for other important covariates such as age, gender, weight, disease stage, performance status, etc. All testing will be 2-sided with a significance level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Priti Tewari, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org